CLINICAL TRIAL: NCT01909791
Title: Treatment for Central-Involved Diabetic Macular Edema in Eyes With Very Good Visual Acuity
Brief Title: Treatment for CI-DME in Eyes With Very Good VA Study
Acronym: Protocol V
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); National Eye Institute (NEI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRCR.net Protocol V; EY14231 (Other Grant/Funding Number: National Eye Institute); EY23207 (Other Grant/Funding Number: National Eye Institute); EY18817 (Other Grant/Funding Number: National Eye Institute)
Record Dates: First submitted 2013-07-23; First posted 2013-07-29 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; anti-vascular endothelial growth factor
MeSH Terms: interventions — Laser Therapy; aflibercept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prompt Laser + Deferred Aflibercept (Experimental): Focal/grid laser followed by intravitreal aflibercept if vision worsens
  Interventions: Procedure: Prompt Laser; Drug: Deferred aflibercept
- Observation + Deferred Aflibercept (Active Comparator): No treatment to start followed by intravitreal aflibercept if vision worsens (deferred laser may be added to intravitreal aflibercept if certain criteria are met)
  Interventions: Procedure: Deferred laser; Drug: Deferred aflibercept
- Prompt Aflibercept (Experimental): Intravitreal aflibercept at baseline and every 4 weeks as needed (deferred laser may be added to intravitreal aflibercept if certain criteria are met)
  Interventions: Drug: Prompt aflibercept; Procedure: Deferred laser

INTERVENTIONS:
Procedure: Prompt Laser — Focal/grid laser performed at baseline and as needed during follow-up
  Other Names: focal/grid photocoagulation; laser treatment
  Arms: Prompt Laser + Deferred Aflibercept
Drug: Prompt aflibercept — Intravitreal injection of 2.0mg aflibercept performed on the day of randomization and up to every 4 weeks using defined treatment criteria
  Other Names: intravitreal anti-VEGF; Eylea
  Arms: Prompt Aflibercept
Procedure: Deferred laser — Focal/grid laser is initiated while receiving anti-VEGF injections only if certain criteria are met
  Other Names: focal/grid photocoagulation; laser treatment
  Arms: Observation + Deferred Aflibercept; Prompt Aflibercept
Drug: Deferred aflibercept — Intravitreal injection of 2.0mg aflibercept performed once certain criteria for vision loss are met and then up to every 4 weeks using defined treatment criteria
  Other Names: intravitreal anti-VEGF; Eylea
  Arms: Observation + Deferred Aflibercept; Prompt Laser + Deferred Aflibercept

SUMMARY:
Although multiple studies have clearly demonstrated that ranibizumab therapy is more effective than laser alone for vision gain and avoiding vision loss in patients with central-involved Diabetic Macular Edema (DME), only eyes with poor visual acuity, such as a visual acuity letter score of 78 or worse (approximate Snellen equivalent of 20/32 or worse) were eligible. Eyes that have central-involved DME with "good" visual acuity (20/25 or better) have not been addressed systematically by recent studies for treatment of DME. Baseline cohort characteristics from the Early Treatment Diabetic Retinopathy Study (ETDRS) suggest that a substantial percentage of eyes with central-involved DME may retain good vision. The investigators do not know definitively whether eyes with central-involved DME and good vision do better with anti-VEGF (vascular endothelial growth factor) (e.g. aflibercept) therapy initially, or focal/grid laser treatment or observation initially followed by anti-VEGF only if vision worsens.

The primary objective of the protocol is to compare the % of eyes that have lost at least 5 letters of visual acuity at 2 years compared with baseline mean visual acuity in eyes with central-involved DME and good visual acuity defined as a Snellen equivalent of 20/25 or better (electronic-ETDRS letter score of 79 or better) that receive (1) prompt focal/grid photocoagulation + deferred anti-VEGF, (2) observation + deferred anti-VEGF, or (3) prompt anti-VEGF.

Secondary objectives include:

* Comparing other visual acuity outcomes between treatment groups, such as the percent of eyes with at least 5, 10 and 15 letter losses in visual acuity from baseline mean visual acuity, percent of eyes with at least 5 letter gain in visual acuity from baseline, mean visual acuity, mean change in visual acuity, adjusted for baseline mean visual acuity
* For eyes randomized to deferred anti-VEGF, the percentage of eyes needing anti-VEGF treatment
* Comparing optical coherence tomography (OCT) outcomes, such as the mean change in OCT central subfield (CSF) thickness, adjusted for baseline mean thickness
* Comparing the number of eyes with PDR at randomization, proportion of eyes avoiding vitreous hemorrhage or panretinal photocoagulation (PRP) or vitrectomy for PDR between treatment groups
* Comparing safety outcomes between treatment groups
* Comparing associated treatment and follow-up exam costs between treatment groups

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Diagnosis of diabetes mellitus (type 1 or type 2)

   Any one of the following will be considered to be sufficient evidence that diabetes is present:
   1. Current regular use of insulin for the treatment of diabetes
   2. Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
   3. Documented diabetes by American Diabetes Association (ADA) and/or World Health Organization (WHO) criteria.
3. Able and willing to provide informed consent.

Meets all of the following ocular criteria in at least the one eye:

1. Best corrected E-ETDRS visual acuity letter score ≥ 79 (approximate Snellen equivalent 20/25 or better) at two consecutive visits within 1 to 28 days.
2. On clinical exam, definite retinal thickening due to DME involving the center of the macula.
3. Diabetic macular edema confirmed on OCT (equivalent to CSF thickness on OCT ≥250 microns on Zeiss Stratus or gender-specific spectral domain OCT equivalent) at two consecutive visits within 1 to 28 days.

   (a) Investigator must verify accuracy of OCT scan by ensuring it is centered and of adequate quality.
4. The investigator is comfortable with the eye being randomized to any of the three treatment groups (observation, laser, or anti-VEGF initially).

   (a) If focal/grid photocoagulation is contraindicated because all leaking microaneurysms are too close to the fovea or the investigator believes the DME that is present will not benefit from focal/grid photocoagulation, the eye should not be enrolled.
5. Media clarity, pupillary dilation, and individual cooperation sufficient for adequate OCT and fundus photographs.

Exclusion Criteria:

1. History of chronic renal failure requiring dialysis or kidney transplant.
2. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
3. Initiation of intensive insulin treatment (a pump or multiple daily injections) within 4 months prior to randomization or plans to do so in the next 4 months.
4. Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval for the indication being studied.

   (a) Note: study participants cannot receive another investigational drug while participating in the study.
5. Known allergy to any component of the study drug.
6. Blood pressure >180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, individual can become eligible.
7. Systemic anti-VEGF or pro-VEGF treatment within 4 months prior to randomization.

   These drugs should not be used during the study.
8. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 24 months.

   (a) Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed.
9. Individual is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the 24 months of the study.

Individual has any of the following ocular characteristics:

1. Macular edema is considered to be due to a cause other than DME.

   a) An eye should not be considered eligible if: (1) the macular edema is considered to be related to ocular surgery such as cataract extraction or (2) clinical exam and/or OCT suggest that vitreoretinal interface abnormalities (e.g., a taut posterior hyaloid or epiretinal membrane) are contributing to the macular edema.
2. An ocular condition is present such that, in the opinion of the investigator, any visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition).
3. An ocular condition is present (other than DME) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.).
4. Cataract is present that, in the opinion of the investigator, may alter visual acuity during the course of the study.
5. Any history of prior laser or other surgical, intravitreal, or peribulbar treatment for DME (such as focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids, or anti-VEGF).
6. History of topical steroid or nonsteroidal anti-inflammatory drugs (NSAID) treatment within 30 days prior to randomization.
7. History of intravitreal or peribulbar corticosteroid within 4 months prior to randomization for an ocular condition other than DME.
8. Any history of or anticipated need for intravitreal anti-VEGF within the next 6 months for an ocular condition other than DME (e.g. choroidal neovascularization, central retinal vein occlusion, PDR).
9. History of PRP within 4 months prior to randomization or anticipated need for PRP in the 6 months following randomization.
10. Any history of vitrectomy.
11. History of major ocular surgery (cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization.
12. History of YAG capsulotomy performed within 2 months prior to randomization.
13. Aphakia.
14. Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2013-10; Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Baker, MD, Study Chair — Paducah Retina Center; Adam Glassman, MS, Principal Investigator — Jaeb Center for Health Research
Locations (103):
- United States (100):
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - University of Arizona Medical Center/Department of Ophthalmology, Tucson, Arizona
  - Jones Eye Institute/University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Retinal Diagnostic Center, Campbell, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - South Coast Retina Center, Long Beach, California
  - Southern California Desert Retina Consultants, MC, Palm Desert, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retinal Consultants of Southern California Medical Group, Inc., Westlake Village, California
  - Retina Group of New England, New London, Connecticut
  - New England Retina Associates, Norwich, Connecticut
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - University of Florida College of Med., Department of Ophthalmology, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Retina Macula Specialists of Miami, Miami, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Ocala Eye Retina Consultants, Ocala, Florida
  - Magruder Eye Institute, Orlando, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Center for Sight, Sarasota, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Retina Associates of Florida, P.A., Tampa, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Glenview, Illinois
  - Illinois Retina Associates, Joliet, Illinois
  - University Retina and Macula Associates, Oak Forest, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Raj Maturi, Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Medical Associates Clinic, P.C., Dubuque, Iowa
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - University of Kansas Medical Center, Dept. of Ophthalmology, Prairie Village, Kansas
  - Retina Associates, P.A., Shawnee Mission, Kansas
  - Retina and Vitreous Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Dept of Ophthalmology and Eye Care Services, Detroit, Michigan
  - Retina Vitreous Center, Grand Blanc, Michigan
  - Retina Specialists of Michigan, Grand Rapids, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Andersen Eye Associates, Saginaw, Michigan
  - Retina Center, PA, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Department of Ophthalmology, Rochester, Minnesota
  - Mid-America Retina Consultants, P.A., Kansas City, Missouri
  - The Retina Institute, St Louis, Missouri
  - Eyesight Ophthalmic Services, PA, Portsmouth, New Hampshire
  - The Institute of Ophthalmology and Visual Science (IOVS), Newark, New Jersey
  - Retinal and Ophthalmic Consultants, PC, Northfield, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Ross Eye Institute, SUNY Buffalo, Buffalo, New York
  - The New York Eye and Ear Infirmary/Faculty Eye Practice, New York, New York
  - MaculaCare, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - University of Rochester, Rochester, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - Western Carolina Retinal Associates, PA, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Oregon Retina, LLP, Eugene, Oregon
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Family Eye Group, Lancaster, Pennsylvania
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania
  - Carolina Retina Center, Columbia, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates, Chattanooga, Tennessee
  - Southeastern Retina Associates, PC, Kingsport, Tennessee
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Southwest Retina Specialists, Amarillo, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Baylor Eye Physicians and Surgeons, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Associates of Utah, P.C., Salt Lake City, Utah
  - Retina Institute of Virginia, Richmond, Virginia
  - Virginia Commonwealth University, Dept. of Ophthalmology, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Spokane Eye Clinic, Spokane, Washington
  - University of Wisconsin-Madison, Dept of Ophthalmology/Retina Service, Madison, Wisconsin
- Canada (3):
  - Alberta Retina Consultants, Edmonton, Alberta
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
  - UBC/VCHA Eye Care Centre, Vancouver

REFERENCES:
- [Background] Glassman AR, Baker CW, Beaulieu WT, Bressler NM, Punjabi OS, Stockdale CR, Wykoff CC, Jampol LM, Sun JK; DRCR Retina Network. Assessment of the DRCR Retina Network Approach to Management With Initial Observation for Eyes With Center-Involved Diabetic Macular Edema and Good Visual Acuity: A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2020 Apr 1;138(4):341-349. doi: 10.1001/jamaophthalmol.2019.6035. PMID 32077907
- [Result] Baker CW, Glassman AR, Beaulieu WT, Antoszyk AN, Browning DJ, Chalam KV, Grover S, Jampol LM, Jhaveri CD, Melia M, Stockdale CR, Martin DF, Sun JK; DRCR Retina Network. Effect of Initial Management With Aflibercept vs Laser Photocoagulation vs Observation on Vision Loss Among Patients With Diabetic Macular Edema Involving the Center of the Macula and Good Visual Acuity: A Randomized Clinical Trial. JAMA. 2019 May 21;321(19):1880-1894. doi: 10.1001/jama.2019.5790. PMID 31037289

RESULTS

PARTICIPANT FLOW:
Groups:
- Initiation With Aflibercept: Intravitreal aflibercept at baseline and every 4 weeks as needed (deferred laser may be added to intravitreal aflibercept if certain criteria are met)
  Prompt aflibercept: Intravitreal injection of 2.0mg aflibercept performed on the day of randomization and up to every 4 weeks using defined treatment criteria
  Deferred laser: Focal/grid laser is initiated while receiving anti-VEGF injections only if certain criteria are met
- Initiation With Laser Photocoagulation: Focal/grid laser followed by intravitreal aflibercept if vision worsens
  Prompt Laser: Focal/grid laser performed at baseline and as needed during follow-up
  Deferred aflibercept: Intravitreal injection of 2.0mg aflibercept performed once certain criteria for vision loss are met and then up to every 4 weeks using defined treatment criteria
- Initiation With Observation: No treatment to start followed by intravitreal aflibercept if vision worsens (deferred laser may be added to intravitreal aflibercept if certain criteria are met)
  Deferred laser: Focal/grid laser is initiated while receiving anti-VEGF injections only if certain criteria are met
  Deferred aflibercept: Intravitreal injection of 2.0mg aflibercept performed once certain criteria for vision loss are met and then up to every 4 weeks using defined treatment criteria
Period: Overall Study
Arm/Group | Initiation With Aflibercept | Initiation With Laser Photocoagulation | Initiation With Observation
Started | 226 | 240 | 236
Completed | 205 | 212 | 208
Not Completed | 21 | 28 | 28
Not completed — Death | 9 | 8 | 4
Not completed — Withdrawal by Subject | 5 | 9 | 13
Not completed — Lost to Follow-up | 5 | 11 | 10
Not completed — Missed Visit | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Initiation With Aflibercept | Initiation With Laser Photocoagulation | Initiation With Observation | Total
Number analyzed (Participants) | 226 | 240 | 236 | 702
Number analyzed (Eyes) | 226 | 240 | 236 | 702
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [52 to 65] | 60 [53 to 66] | 60 [53 to 67] | 60 [52 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 82 | 87 | 264
  Male | 131 | 158 | 149 | 438
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic White | 145 | 160 | 161 | 466
  Race/ethnicity: Non-Hispanic Black/African American | 37 | 36 | 41 | 114
  Race/ethnicity: Hispanic or Latino | 31 | 35 | 25 | 91
  Race/ethnicity: Asian | 6 | 1 | 5 | 12
  Race/ethnicity: American Indian or Alaskan Native | 1 | 1 | 0 | 2
  Race/ethnicity: Native Hawaiian or other Pacific Islander | 0 | 3 | 1 | 4
  Race/ethnicity: More than one race | 4 | 2 | 1 | 7
  Race/ethnicity: Unknown or not reported | 2 | 2 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1 | 2 | 4 | 7
  United States | 225 | 238 | 232 | 695
Diabetes type [Count of Participants; unit: Participants]
  Type 2 | 211 | 221 | 210 | 642
  Type 1 | 13 | 18 | 18 | 49
  Uncertain | 2 | 1 | 8 | 11
Duration of diabetes [Median (Inter-Quartile Range); unit: years] | 15 [10 to 21] | 15 [10 to 20] | 16 [10 to 24] | 15 [10 to 21]
Insulin used [Count of Participants; unit: Participants] | 161 | 145 | 160 | 466
Hemoglobin A1c [Median (Inter-Quartile Range); unit: Hemoglobin A1c percentage] — Population: Hemoglobin A1c was missing for 9,8, and 10 eyes in the initiation with aflibercept, initiation with laser photocoagulation, and initiation with observation groups, respectively.
  Hemoglobin A1c percentage
    number analyzed (Participants) | 217 | 232 | 226 | 675
    (all) | 7.6 [6.8 to 9.1] | 7.6 [6.6 to 8.6] | 7.6 [6.8 to 8.7] | 7.6 [6.7 to 8.8]
Arterial blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 99 [91 to 107] | 98 [89 to 105] | 98 [91 to 105] | 98 [90 to 106]
Prior myocardial infarction [Count of Participants; unit: Participants] | 11 | 21 | 19 | 51
Prior stroke [Count of Participants; unit: Participants] | 16 | 6 | 9 | 31
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] — Calculated as weight in kilograms divided by height in meters squared Population: Missing for 42, 33, and 37 participants in the aflibercept, laser and observation groups, respectively.
  kg/m^2
    number analyzed (Participants) | 184 | 207 | 199 | 590
    (all) | 32.3 [27.6 to 37.0] | 32.1 [28.2 to 37.4] | 32.3 [28.0 to 37.5] | 32.2 [28.0 to 37.3]
Daily cigarette smoking [Count of Participants; unit: Participants]
  Never | 165 | 157 | 141 | 463
  Prior | 46 | 67 | 75 | 188
  Current | 15 | 16 | 20 | 51
Recent or planned diabetic macular edema treatment in non-study eye [Count of Units; unit: Eyes] | 86 | 90 | 92 | 268
Prior treatment for diabetic macular edema [Count of Units; unit: Eyes] | 34 | 31 | 34 | 99
Prior anti-VEGF for diabetic macular edema [Count of Units; unit: Eyes] | 11 | 14 | 13 | 38
Prior focal/grid laser photocoagulation for diabetic macular edema [Count of Units; unit: Eyes] | 26 | 24 | 24 | 74
Prior panretinal photocoagulation [Count of Units; unit: Eyes] | 15 | 12 | 9 | 36
Lens status at clinical examination [Count of Units; unit: Eyes]
  Phakic (natural lens) | 180 | 188 | 182 | 550
  Prosthetic intraocular lens | 46 | 52 | 54 | 152
E-ETDRS visual acuity letter score [Mean (Standard Deviation); unit: units on a scale] — Average of screening and randomization values. Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/12) to 0 letters (Snellen equivalent of 20/800).
  units on a scale | 85.2 (3.5) | 85.2 (3.8) | 85.2 (3.8) | 85.2 (3.7)
Intraocular pressure [Median (Inter-Quartile Range); unit: mmHg] | 15 [13 to 18] | 15 [13 to 18] | 15 [13 to 18] | 15 [13 to 18]
Patient-reported visual complaints presumed to be from diabetic macular edema [Count of Units; unit: Eyes] | 99 | 116 | 118 | 333
Optical coherence tomography machine used to measure central subfield thickness [Count of Units; unit: Eyes] — An optical coherence tomography machine is the device that was used to measure the central subfield thickness.
  Eyes
    Heidelberg Spectralis | 148 | 151 | 151 | 450
    Zeiss Cirrus | 78 | 89 | 85 | 252
Central subfield thickness (time-domain equivalent) [Mean (Standard Deviation); unit: Microns] — Calculated as the average of screening and randomization values.
  Microns | 306 (55) | 314 (52) | 314 (64) | 311 (57)
Macular volume (time-domain equivalent) [Mean (Standard Deviation); unit: mm^3] — Average of screening and randomization values. Population: missing for one participant in the observation group
  mm^3
    number analyzed (Participants) | 226 | 240 | 236 | 701
    number analyzed (Eyes) | 226 | 240 | 235 | 701
    (all) | 7.9 (1.1) | 8.0 (1.2) | 8.0 (1.1) | 8.0 (1.0)
Diabetic retinopathy severity level [Count of Units; unit: Eyes] — Graded by a central reading center. PDR, proliferative diabetic retinopathy, NPDR, non-proliferative diabetic retinopathy Population: Missing for 10, 13, and 7 eyes in the aflibercept, laser, and observation groups, respectively.
  Eyes
    number analyzed (Eyes) | 216 | 227 | 229 | 672
    Diabetic Retinopathy absent or questionable | 2 | 4 | 1 | 7
    Microaneurysms only | 13 | 8 | 6 | 27
    Mild to moderate NPDR | 119 | 132 | 142 | 393
    Moderately severe to severe NPDR | 58 | 64 | 62 | 184
    Inactive PDR | 6 | 7 | 7 | 20
    Mild to moderate PDR | 14 | 12 | 9 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With at Least 5-letter Decrease in E-ETDRS Visual Acuity Letter Score From Baseline
Description: Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/12) to 0 letters (Snellen equivalent of 20/800).
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Initiation With Aflibercept | Initiation With Laser Photocoagulation | Initiation With Observation
Number analyzed (Participants) | 205 | 212 | 208
Number analyzed (Eyes) | 205 | 212 | 208
Eyes | 33 | 36 | 39

2. Secondary Outcome: Number of Eyes With at Least 5-letter Increase or at Least 5-, 10-, or 15-letter Decrease in E-ETDRS Visual Acuity Letter Score From Baseline
Description: as for outcome 1
Time Frame: 1 year
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Initiation With Aflibercept | Initiation With Laser Photocoagulation | Initiation With Observation
Number analyzed (Participants) | 210 | 226 | 220
Number analyzed (Eyes) | 210 | 226 | 220
Eyes
  ≥ 5-Letter Increase | 61 | 44 | 33
  ≥ 5-Letter Decrease | 19 | 36 | 25
  ≥ 10-Letter Decrease | 6 | 9 | 7
  ≥ 15-Letter Decrease | 3 | 4 | 6

3. Secondary Outcome: Change in E-ETDRS Visual Acuity Letter Score From Baseline
Description: as for outcome 1
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Initiation With Aflibercept | Initiation With Laser Photocoagulation | Initiation With Observation
Number analyzed (Participants) | 210 | 226 | 220
Number analyzed (Eyes) | 210 | 226 | 220
units on a scale | 2.1 (5.0) | 0.1 (5.5) | 0.0 (5.4)

4. Secondary Outcome: Change in E-ETDRS Visual Acuity Letter Score From Baseline Over 2 Years (Area Under the Curve)
Description: Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/12) to 0 letters (Snellen equivalent of 20/800). The area under the curve (units = letters·years) was divided by 2 years (units = years) to obtain an average change in letter score (units = letters) over the 2-year follow-up.
Time Frame: 2 year
Population: Best-corrected visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the early treatment diabetic retinopathy study method . Best value on the scale 100, worst 0.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Initial Aflibercept: Intravitreal aflibercept at baseline and every 4 weeks as needed (deferred laser may be added to intravitreal aflibercept if certain criteria are met)
  Prompt aflibercept: Intravitreal injection of 2.0mg aflibercept performed on the day of randomization and up to every 4 weeks using defined treatment criteria
  Deferred laser: Focal/grid laser is initiated while receiving anti-VEGF injections only if certain criteria are met
- Initial Laser With Deferred Aflibercept if Needed: Focal/grid laser followed by intravitreal aflibercept if vision worsens
  Prompt Laser: Focal/grid laser performed at baseline and as needed during follow-up
  Deferred aflibercept: Intravitreal injection of 2.0mg aflibercept performed once certain criteria for vision loss are met and then up to every 4 weeks using defined treatment criteria
- Observation: No treatment to start followed by intravitreal aflibercept if vision worsens (deferred laser may be added to intravitreal aflibercept if certain criteria are met)
  Deferred laser: Focal/grid laser is initiated while receiving anti-VEGF injections only if certain criteria are met
  Deferred aflibercept: Intravitreal injection of 2.0mg aflibercept performed once certain criteria for vision loss are met and then up to every 4 weeks using defined treatment criteria
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 205 | 212 | 208
Number analyzed (Eyes) | 205 | 212 | 208
units on a scale | 1.5 (4.0) | 0.0 (3.9) | -0.4 (4.2)

5. Secondary Outcome: Change in OCT Central Subfield Thickness From Baseline
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 205 | 212 | 207
Number analyzed (Eyes) | 205 | 212 | 207
microns | -48 (65) | -41 (75) | -42 (75)

6. Secondary Outcome: Number of Eyes With at Least 1 or 2 Logarithmic-step Central Subfield Thickness Improvement and Worsening
Description: Logarithmic transformation of optical coherence tomography central subfield thickness (CST) is calculated by taking the log base 10 of the ratio of the central subfield thickness divided by 200 and rounding to the nearest hundredth. The change is the change in the log values.
Time Frame: 1 year
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 210 | 223 | 220
Number analyzed (Eyes) | 210 | 223 | 220
Eyes
  ≥ 2 log-step CST decrease (improvement) | 7 | 11 | 8
  ≥ 1 log-step CST decrease (improvement) | 56 | 45 | 39
  ≥ 1 log-step CST increase (worsening) | 1 | 12 | 14
  ≥ 2 log-step CST increase (worsening) | 0 | 3 | 3

7. Secondary Outcome: Number of Eyes With no Center-involved Diabetic Macular Edema and at Least 10% Central Subfield Thickness Decrease
Description: Center-involved diabetic macular edema defined as follows by central subfield thickness according to optical coherence tomography machine and sex: Heidelberg Spectralis ≥ 305 µm in women and ≥ 320 µm in men, and Zeiss Cirrus ≥ 290 µm in women and ≥ 305 µm in men.
Time Frame: 1 year
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 210 | 223 | 220
Number analyzed (Eyes) | 210 | 223 | 220
Eyes | 93 | 58 | 67

8. Secondary Outcome: Cumulative Number of Intraocular Injections of 2.0-mg Aflibercept Received Per Participant
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Injections
Units Other Than Participants: Eyes
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 210 | 226 | 220
Number analyzed (Eyes) | 210 | 226 | 220
Injections | 6.0 (2.5) | 0.7 (2.1) | 1.4 (2.6)

9. Secondary Outcome: Number of Eyes With ≥ 2-step Worsening of Diabetic Retinopathy
Description: Includes eyes with baseline severity level of 75 (high-risk proliferative diabetic retinopathy) or less based on reading center grading of color fundus photographs using the Early Treatment Diabetic Retinopathy Study severity scale.
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 185 | 187 | 188
Number analyzed (Eyes) | 185 | 187 | 188
Eyes | 7 | 18 | 20

10. Secondary Outcome: For Eyes Randomized to Initial Laser Photocoagulation and Initial Observation Groups, the Percentage Receiving Aflibercept Treatment
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Initiation With Laser Photocoagulation | Initiation With Observation
Number analyzed (Participants) | 240 | 236
Number analyzed (Eyes) | 240 | 236
Eyes | 60 | 80

11. Secondary Outcome: Number of Eyes With at Least 5-, 10-, or 15-letter Decrease in E-ETDRS Visual Acuity Letter Score From Baseline
Description: as for outcome 1
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Initiation With Aflibercept | Initiation With Laser Photocoagulation | Initiation With Observation
Number analyzed (Participants) | 205 | 212 | 208
Number analyzed (Eyes) | 205 | 212 | 208
Eyes
  ≥ 5-Letter Improvement | 55 | 53 | 43
  ≥ 10-Letter Worsening | 18 | 14 | 14
  ≥ 15-Letter Worsening | 5 | 8 | 8

12. Secondary Outcome: Change in E-ETDRS Visual Acuity Letter Score From Baseline
Description: as for outcome 1
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Initiation With Aflibercept | Initiation With Laser Photocoagulation | Initiation With Observation
Number analyzed (Participants) | 205 | 212 | 208
Number analyzed (Eyes) | 205 | 212 | 208
units on a scale | 0.9 (6.4) | 0.1 (6.3) | -0.4 (6.4)

13. Secondary Outcome: Change in OCT Central Subfield Thickness From Baseline
Description: Measured using spectral-domain optical coherence tomography (OCT).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 210 | 223 | 220
Number analyzed (Eyes) | 210 | 223 | 220
microns | -50 (55) | -30 (69) | -25 (73)

14. Secondary Outcome: Number of Eyes With at Least 1 or 2 Logarithmic-step Central Subfield Thickness Improvement and Worsening
Description: Logarithmic transformation of optical coherence tomography central subfield thickness is calculated by taking the log base 10 of the ratio of the central subfield thickness divided by 200 and rounding to the nearest hundredth. The change is the change in the log values.
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 205 | 212 | 207
Number analyzed (Eyes) | 205 | 212 | 207
Eyes
  ≥ 2 log-step CST decrease (improvement) | 12 | 18 | 13
  ≥ 1 log-step CST decrease (improvement) | 57 | 56 | 61
  ≥ 1 log-step CST increase (worsening) | 6 | 10 | 11
  ≥ 2 log-step CST increase (worsening) | 1 | 1 | 2

15. Secondary Outcome: Number of Eyes With no Center-involved Diabetic Macular Edema and at Least 10% Central Subfield Thickness Decrease
Description: as for outcome 7
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 205 | 212 | 207
Number analyzed (Eyes) | 205 | 212 | 207
Eyes | 95 | 90 | 74

16. Secondary Outcome: Cumulative Number of Focal/Grid Photocoagulation Sessions Performed Per Participant
Time Frame: 2 years
Population: The initial laser session was completed for all eyes in the initial laser group.
Measure: Mean (Standard Deviation); unit: Focal/grid photocoagulation session
Units Other Than Participants: Eyes
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 205 | 212 | 208
Number analyzed (Eyes) | 205 | 212 | 208
Focal/grid photocoagulation session | 0.1 (0.4) | 1.5 (0.9) | 0.0 (0.3)

17. Secondary Outcome: Number of Eyes With ≥ 2-step Improvement of Diabetic Retinopathy
Description: Includes eyes with baseline severity level of 35 (mild non-proliferative diabetic retinopathy) or greater based on reading center grading of color fundus photographs using the Early Treatment Diabetic Retinopathy Study severity scale. Excludes eyes with severity level 60 at baseline since improvement is not possible in these eyes.
Time Frame: 2 years
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 165 | 170 | 177
Number analyzed (Eyes) | 165 | 170 | 177
Eyes | 23 | 21 | 18

18. Secondary Outcome: Cumulative Number of Intraocular Injections of 2.0-mg Aflibercept Received Per Participant
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Injections
Units Other Than Participants: Eyes
Arm/Group | Initial Aflibercept | Initial Laser With Deferred Aflibercept if Needed | Observation
Number analyzed (Participants) | 205 | 212 | 208
Number analyzed (Eyes) | 205 | 212 | 208
Injections | 8.3 (4.2) | 2.1 (4.0) | 3.1 (4.9)

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Initiation With Laser Photocoagulation | Initiation With Observation | Initiation With Aflibercept
All-Cause Mortality (participants affected / at risk) | 10/226 | 9/240 | 5/236
Serious Adverse Events (participants affected / at risk) | 64/240 | 77/236 | 69/226
Other Adverse Events (participants affected / at risk) | 194/240 | 197/236 | 185/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initiation With Laser Photocoagulation (N=240) | Initiation With Observation (N=236) | Initiation With Aflibercept (N=226)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Bicuspid aortic valve (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (3) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (6) | 5 (5) | 5 (5)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3) | 5 (5)
Diabetes mellitus inadequate control (Endocrine disorders) | 0 (0) | 2 (3) | 2 (2)
Diabetic coma (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Endocrine disorders) | 1 (1) | 3 (3) | 0 (0)
Hyperglycaemia (Endocrine disorders) | 1 (1) | 1 (1) | 2 (2)
Hypoglycaemia (Endocrine disorders) | 0 (0) | 1 (1) | 2 (2)
Thyroid cancer (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract traumatic (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 4 (4) | 6 (7) | 3 (3)
Death (General disorders) | 3 (3) | 2 (2) | 3 (3)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Flank pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (4) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 4 (4) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood electrolytes decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Lower limb fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Multiple fractures (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0)
Cardiorenal syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (2) | 1 (1) | 2 (2)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 4 (4) | 1 (1) | 1 (1)
Breast cancer (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 6 (7)
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cardiac operation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel decompression (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 1 (1) | 2 (2)
Gastric banding (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 3 (3)
Knee operation (Surgical and medical procedures) | 1 (1) | 1 (1) | 3 (3)
Leg amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Stent placement (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Surgery (Surgical and medical procedures) | 3 (3) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1)
Vascular graft (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery disease (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Cerebral haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 5 (5) | 3 (3) | 3 (3)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Ischaemic stroke (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initiation With Laser Photocoagulation (N=240) | Initiation With Observation (N=236) | Initiation With Aflibercept (N=226)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 9 (9) | 4 (4)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 3 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 5 (6) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 4 (4) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Long QT syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 4 (4) | 5 (5) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Mastoiditis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Endocrine disorders) | 9 (11) | 8 (8) | 4 (5)
Diabetes mellitus inadequate control (Endocrine disorders) | 9 (10) | 7 (8) | 7 (7)
Diabetic ketoacidosis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Endocrine disorders) | 2 (2) | 1 (1) | 2 (2)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Endocrine disorders) | 2 (2) | 0 (0) | 4 (6)
Hypothyroidism (Endocrine disorders) | 0 (0) | 6 (6) | 2 (2)
Pituitary tumour benign (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroid neoplasm (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3)
Age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Altered visual depth perception (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenopia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 2 (3) | 3 (3) | 1 (1)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Borderline glaucoma (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 14 (14) | 14 (15) | 17 (17)
Cataract cortical (Eye disorders) | 6 (6) | 6 (6) | 11 (11)
Cataract nuclear (Eye disorders) | 4 (4) | 1 (1) | 8 (8)
Cataract subcapsular (Eye disorders) | 4 (4) | 4 (6) | 11 (13)
Chalazion (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 8 (11) | 9 (13) | 17 (23)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 3 (3) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 1 (1) | 2 (2)
Conjunctivitis viral (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Corneal abrasion (Eye disorders) | 2 (2) | 2 (3) | 3 (4)
Corneal defect (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Corneal disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal dystrophy (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Corneal erosion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Corneal oedema (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Corneal opacity (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Corneal pigmentation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal scar (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cystoid macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinal oedema (Eye disorders) | 6 (6) | 7 (7) | 2 (2)
Diabetic retinopathy (Eye disorders) | 6 (7) | 2 (2) | 5 (5)
Diplopia (Eye disorders) | 8 (8) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 11 (12) | 8 (10) | 17 (18)
Eye discharge (Eye disorders) | 1 (1) | 2 (2) | 1 (1)
Eye irritation (Eye disorders) | 6 (6) | 7 (7) | 12 (13)
Eye pain (Eye disorders) | 5 (8) | 11 (14) | 16 (19)
Eye pruritus (Eye disorders) | 9 (10) | 3 (3) | 6 (6)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eyelid margin crusting (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Eyelid pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Foreign body in eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 2 (3) | 3 (3) | 2 (2)
Glare (Eye disorders) | 6 (6) | 1 (1) | 0 (0)
Hordeolum (Eye disorders) | 5 (5) | 2 (2) | 1 (2)
Hyalosis asteroid (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hyphaema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Iris adhesions (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Iris neovascularisation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 9 (9) | 8 (10) | 8 (8)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 10 (10) | 1 (1) | 6 (7)
Macular ischaemia (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Macular oedema (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Meibomian gland dysfunction (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Metamorphopsia (Eye disorders) | 3 (3) | 2 (2) | 3 (4)
Ocular discomfort (Eye disorders) | 3 (3) | 3 (4) | 7 (7)
Ocular hyperaemia (Eye disorders) | 0 (0) | 3 (3) | 6 (6)
Ocular hypertension (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Ophthalmic herpes simplex (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Optic atrophy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Optic nerve cupping (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 4 (4) | 7 (8) | 8 (8)
Photopsia (Eye disorders) | 3 (3) | 4 (4) | 7 (7)
Posterior capsule opacification (Eye disorders) | 3 (3) | 1 (1) | 2 (2)
Punctate keratitis (Eye disorders) | 3 (3) | 2 (3) | 4 (4)
Retinal aneurysm (Eye disorders) | 3 (3) | 5 (5) | 3 (3)
Retinal artery embolism (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal exudates (Eye disorders) | 5 (6) | 12 (12) | 7 (7)
Retinal haemorrhage (Eye disorders) | 2 (2) | 10 (11) | 4 (4)
Retinal ischaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal neovascularisation (Eye disorders) | 5 (5) | 3 (3) | 2 (3)
Retinal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal pigment epitheliopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 2 (2) | 2 (2) | 1 (1)
Retinal vein occlusion (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Retinopathy hypertensive (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Subretinal fibrosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 31 (39) | 34 (43) | 40 (46)
Visual acuity reduced (Eye disorders) | 15 (16) | 16 (16) | 6 (6)
Visual field defect (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 11 (12) | 11 (13) | 9 (11)
Vitreous adhesions (Eye disorders) | 0 (0) | 3 (3) | 2 (2)
Vitreous detachment (Eye disorders) | 3 (3) | 4 (4) | 12 (12)
Vitreous disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 16 (16) | 21 (22) | 27 (34)
Vitreous haemorrhage (Eye disorders) | 6 (7) | 5 (5) | 8 (11)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (4) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 6 (6) | 8 (9)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Gastroenteritis viral (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 6 (6) | 7 (7)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 11 (12) | 8 (9) | 7 (8)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Tooth fracture (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Tooth infection (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (5)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (3) | 0 (0) | 6 (7)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (4) | 7 (8)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 1 (1)
Chest pain (General disorders) | 4 (4) | 7 (7) | 3 (4)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 4 (4) | 5 (5)
Flank pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (General disorders) | 0 (0) | 2 (2) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (2) | 0 (0)
Necrosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 8 (10) | 8 (8) | 3 (3)
Pain (General disorders) | 3 (3) | 2 (2) | 4 (5)
Peripheral swelling (General disorders) | 1 (1) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 6 (6)
Swelling (General disorders) | 2 (2) | 3 (3) | 4 (4)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 2 (2)
Seasonal allergy (Immune system disorders) | 7 (7) | 2 (2) | 6 (6)
Systemic lupus erythematosus (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Urticaria (Immune system disorders) | 0 (0) | 3 (3) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 4 (4) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 7 (7) | 9 (10) | 10 (11)
Localised infection (Infections and infestations) | 3 (3) | 2 (2) | 8 (10)
Onychomycosis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Streptococcal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 5 (5)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chemical injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 5 (8) | 4 (4)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (2) | 2 (2) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 4 (4)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (4)
Biopsy skin (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood testosterone decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Carotid bruit (Investigations) | 0 (0) | 0 (0) | 1 (1)
Echocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Free prostate-specific antigen increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 1 (1) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 2 (2) | 1 (1) | 3 (3)
Laboratory test abnormal (Investigations) | 0 (0) | 2 (9) | 2 (3)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 (5) | 5 (5) | 7 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3) | 8 (8) | 3 (3)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 10 (11) | 7 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5) | 3 (3)
Arthritis bacterial (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 8 (8) | 9 (10)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Foot fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Hand fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Joint dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Lipoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Multiple fractures (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 2 (2)
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (6) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 3 (4)
Myokymia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 11 (14) | 10 (10)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Stiff person syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (8)
Wrist fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 0 (0)
Apraxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Benign intracranial hypertension (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 2 (3) | 2 (2) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 7 (7) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 7 (8) | 7 (8)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (8) | 14 (16) | 15 (17)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 4 (5) | 1 (1) | 5 (5)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Nerve injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 5 (5) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ulnar nerve injury (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 7 (7) | 6 (7) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (4) | 6 (6) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 5 (5) | 3 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3) | 3 (3)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 5 (5) | 5 (5) | 1 (1)
Cystitis (Renal and urinary disorders) | 3 (3) | 2 (2) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (3) | 2 (2) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3)
Kidney infection (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (3) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 5 (5) | 3 (3) | 2 (2)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 13 (17) | 5 (6) | 6 (8)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 0 (0) | 4 (6)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 16 (19) | 9 (10)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (9) | 8 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 15 (16) | 23 (26)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 5 (5) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 13 (20) | 10 (10) | 7 (7)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 3 (3)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 12 (13) | 8 (9)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 2 (4) | 4 (4) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Cellulitis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 6 (6)
Contusion (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Cutis laxa (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Dermatophytosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 5 (5)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Herpes zoster (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Nail avulsion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Onychogryphosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 4 (4)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin bacterial infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin cancer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Arterial bypass operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Benign tumour excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Bile duct stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Blepharoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 2 (2) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Dental implantation (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 2 (2) | 2 (2)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 2 (3) | 1 (1) | 0 (0)
Metatarsal excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Retinal laser coagulation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Skin graft (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Skin lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Stent placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 2 (2) | 3 (3)
Transfusion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Wrist surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1) | 1 (2)
Carotid artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 20 (20) | 18 (20) | 13 (13)
Hypotension (Vascular disorders) | 3 (3) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Transient ischaemic attack (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-04-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT01909791/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT01909791/SAP_001.pdf